CLINICAL TRIAL: NCT03596528
Title: Interstitial Lung Disease (ILD). Comparative Study of the Diagnostic Yield of Surgical Lung Biopsy Versus Cryobiopsy.
Brief Title: Interstitial Lung Disease (ILD). Diagnostic Yield of Surgical Lung Biopsy Versus Cryobiopsy in the Same Surgical Stage.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Alejandra Libreros Niño, MD, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCB/2017/0900
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Lung Diseases, Interstitial
Keywords: Interstitial lung disease, cryobiopsy, surgical biopsy
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung biopsy (Other): Lung biopsy
  Interventions: Procedure: Lung biopsy

INTERVENTIONS:
Procedure: Lung biopsy — Each patient will be brought to the operating room and will undergo cryobiopsy and surgical biopsy of the lung sequentially in the same surgical stage.
  Other Names: Cryobiopsy

SUMMARY:
In patients with interstitial lung disease (ILD) with inconsistent clinical and radiological features, establishing a reliable diagnosis of ILD requires a surgical lung biopsy

Transbronchial cryobiopsy is a minimally invasive, rapid, safe technique, and with histologic diagnostic yields, for ILD, typically exceeding 70 -80% .

The aim of this study is to compare and analyze the diagnostic yield, for ILD, and complications following SLB and TC

Methods. The investigators designed a descriptive, comparative and cross-sectional study in patients with ILD, in which SLB and CT will be performed in the same surgical stage, as diagnostic tests.

This study will be conducted from January 2018 to January 2019. Surgical lung biopsy and TC will be performed in the same surgical stage in all patients, under general anesthesia and mechanical ventilation. First TC will be performed by a pulmonologist, sequentially a thoracic surgeon will carry out a SLB.

The samples obtained will be analyzed by different pathologist to compare both techniques in terms of histologic features.

Diagnostic yield, postoperative complications, comorbidities and lenght of stay will be analyzed and compared following these procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients for suspected ILD eligible for lung biopsy reviewed during multidisciplinary approach.
* Subject provides informed consent.
* A negative pregnancy test in women of child-bearing potential.
* Subject is mentally capable of understanding study procedures.
* 18 years and older.

Exclusion Criteria:

* Study subject has any disease or condition that interferes with safe completion of the study including:
* Platelet count < 50,000 or Coagulopathy defined as an International Normalized Ratio (INR) > 1.5 on the day of procedure, as well as discontinuation of ticagrelor or clopidogrel within 5 days of procedure.
* Severely impaired lung function as determined with spirometry evidenced by a forced expiratory volume in 1 second (FEV1) < 0.8, or radiographically as diffuse bullous disease
* Hemodynamic instability with systolic blood pressure <90 mmHg or heart rate > 120 beats/min, unless deemed to be stable with these values by the surgical or interventional pulmonary attending physicians
* Hypoxemia with pulse oximetry values <88% or partial pressure of oxygen in arterial blood (PaO2) < 60 on baseline oxygen requirements
* Concurrent participation in another study involving investigational drugs or investigational medical devices
* Inability to read and understand the necessary study documents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03-23 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of the tissue sample reported by the pathologist. | for statistical analysis, 12 months after the first inclusion
  comparison of diagnostic yield of cryobiopsy versus surgical lung biopsy according to the quality of the tissue sample reported by the pathologist.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Background] Xaubet A, Ancochea J, Bollo E, Fernandez-Fabrellas E, Franquet T, Molina-Molina M, Montero MA, Serrano-Mollar A; Sociedad Espanola de Neumologia y Cirugia Toracica (SEPAR) Research Group on Diffuse Pulmonary Diseases. Guidelines for the diagnosis and treatment of idiopathic pulmonary fibrosis. Sociedad Espanola de Neumologia y Cirugia Toracica (SEPAR) Research Group on Diffuse Pulmonary Diseases. Arch Bronconeumol. 2013 Aug;49(8):343-53. doi: 10.1016/j.arbres.2013.03.011. Epub 2013 Jun 4. English, Spanish. PMID 23742884
- [Background] Walker CM, Chung JH, Wall C, Pipavath SN, Chapman T, Reddy GP, Stern EJ, Godwin JD, Weinberger E. Interactive high-resolution computed tomography digital atlas of interstitial lung disease. Acad Radiol. 2011 Nov;18(11):1453-60. doi: 10.1016/j.acra.2011.07.008. Epub 2011 Sep 1. PMID 21889896
- [Background] Rena O, Casadio C, Leo F, Giobbe R, Cianci R, Baldi S, Rapellino M, Maggi G. Videothoracoscopic lung biopsy in the diagnosis of interstitial lung disease. Eur J Cardiothorac Surg. 1999 Dec;16(6):624-7. doi: 10.1016/s1010-7940(99)00320-6. PMID 10647831
- [Background] American Thoracic Society. Idiopathic pulmonary fibrosis: diagnosis and treatment. International consensus statement. American Thoracic Society (ATS), and the European Respiratory Society (ERS). Am J Respir Crit Care Med. 2000 Feb;161(2 Pt 1):646-64. doi: 10.1164/ajrccm.161.2.ats3-00. No abstract available. PMID 10673212
- [Background] Lentz RJ, Argento AC, Colby TV, Rickman OB, Maldonado F. Transbronchial cryobiopsy for diffuse parenchymal lung disease: a state-of-the-art review of procedural techniques, current evidence, and future challenges. J Thorac Dis. 2017 Jul;9(7):2186-2203. doi: 10.21037/jtd.2017.06.96. PMID 28840020
- [Background] Fibla JJ, Molins L, Simon C, Perez J, Vidal G. Early removal of chest drainage after videothoracoscopic lung biopsy. Interact Cardiovasc Thorac Surg. 2006 Oct;5(5):581-3. doi: 10.1510/icvts.2006.129338. Epub 2006 Jun 28. PMID 17670651
- [Background] Katzenstein AL, Myers JL. Idiopathic pulmonary fibrosis: clinical relevance of pathologic classification. Am J Respir Crit Care Med. 1998 Apr;157(4 Pt 1):1301-15. doi: 10.1164/ajrccm.157.4.9707039. No abstract available. PMID 9563754
- [Background] Hodnett PA, Naidich DP. Fibrosing interstitial lung disease. A practical high-resolution computed tomography-based approach to diagnosis and management and a review of the literature. Am J Respir Crit Care Med. 2013 Jul 15;188(2):141-9. doi: 10.1164/rccm.201208-1544CI. PMID 23672718
- [Background] Shorr AF, Lettieri CJ, Helman DL. Role for transbronchial biopsy in the diagnosis of usual interstitial pneumonia. Chest. 2007 Jan;131(1):329-30; author reply 330. doi: 10.1378/chest.06-1266. No abstract available. PMID 17218598
- [Background] Babiak A, Hetzel J, Krishna G, Fritz P, Moeller P, Balli T, Hetzel M. Transbronchial cryobiopsy: a new tool for lung biopsies. Respiration. 2009;78(2):203-8. doi: 10.1159/000203987. Epub 2009 Feb 21. PMID 19246874
- [Background] Berbescu EA, Katzenstein AL, Snow JL, Zisman DA. Transbronchial biopsy in usual interstitial pneumonia. Chest. 2006 May;129(5):1126-31. doi: 10.1378/chest.129.5.1126. PMID 16685001
- [Result] Xaubet A, Ancochea J, Blanquer R, Montero C, Morell F, Rodriguez Becerra E, Sueiro A, Villena V; Grupo de Investigacion en Enfermedades Pulmonares Intersticiales Difusas. Area de Tecnicas y Transplante. SEPAR. [Diagnosis and treatment of diffuse interstitial lung diseases]. Arch Bronconeumol. 2003 Dec;39(12):580-600. doi: 10.1016/s0300-2896(03)75457-x. No abstract available. Spanish. PMID 14636495